CLINICAL TRIAL: NCT03865121
Title: Uncontrolled Pilot Trial of Transnasal Nicotine in Parkinson Disease
Brief Title: Pilot Trial of Transnasal Nicotine in Parkinson Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Collaborators: Howard University (Other)
Responsible Party: Principal Investigator, Leo Bayliss-Amaya, Attending Neurologist, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNNMVS
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Nicotine; Transnasal
MeSH Terms: conditions — Parkinson Disease | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Uncontrolled Pilot Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nicotine Nasal Spray 10 MG/ML (Experimental): Patients will receive incremental doses of Nicotine Nasal Spray 10 MG/ML (0.5 MG/SPRAY) starting with 3 bilateral puffs per day (3 mg total) for 3 days, followed by 5 bilateral puffs per day (5 mg) for 3 days, followed by 8 bilateral puffs per day (8 mg) for 4 days, followed by 10 bilateral puffs per day (10 mg) for 10 days.
  Interventions: Drug: Nicotine Nasal Spray 10 MG/ML (0.5 MG/SPRAY)

INTERVENTIONS:
Drug: Nicotine Nasal Spray 10 MG/ML (0.5 MG/SPRAY) — Patients will receive incremental doses of Nicotine Nasal Spray 10 MG/ML (0.5 MG/SPRAY) starting with 3 bilateral puffs per day (3 mg total) for 3 days, followed by 5 bilateral puffs per day (5 mg) for 3 days, followed by 8 bilateral puffs per day (8 mg) for 4 days, followed by 10 bilateral puffs per day (10 mg) for 10 days.
  Other Names: Nicotine Nasal Spray

SUMMARY:
The widely observed inverse relationship between smoking and Parkinson's Disease (PD) and the results of numerous preclinical studies indicating neuroprotective effects of nicotine, suggest a possible novel intervention in PD. In our opinion, an optimal nicotinic therapy in PD would consist of pulsatile nicotine delivery (e.g. via nasal spray) similar to pulsatile nicotine obtained via smoking. The investigators believe that pulsatile stimulation of the central nicotinic receptors (achievable via nasal spray) would affect the dynamic of the nicotinic receptors much more desirably and similar to smoking compared to continuous nicotine administration via patch, which might result in continuous nicotinic receptor desensitization. Thus, this pilot trial seeks to evaluate the efficacy of nicotine nasal spray (Nicotrol NS®) in symptomatology of PD. For this purpose, a total of 6 non-smoking patients at intermediate disease stages (2-3 of Hoehn and Yahr scale) and receiving conventional therapy for PD will be recruited at the "Instituto Nacional de Neurología y Neurocirugía, (Manuel Velasco Suárez)" in Mexico City. Nicotrol NS® in incremental dosing (up to 10 mg/day) regimens will be added to the current medications to each patient during the first week. This will be maintained for up to 1 month. Motor and non-motor aspects of PD will be evaluated. The investigators expect significant improvement of motor and non-motor symptoms in all patients receiving Nicotrol NS® during therapy and a reversal during withdrawal.

DETAILED DESCRIPTION:
Parkinson's disease (PD), the second most common progressive neurodegenerative disorder, is associated with loss of dopaminergic neurons in the substantia nigra pars compacta that leads to striatal dopamine deficiency. This dopaminergic loss results in motor deficits characterized by: akinesia, rigidity, resting tremor and postural instability as well as non-motor symptoms that might also involve other neurotransmitter systems. The non-motor symptoms may include: cognitive deficits (e.g., mild to severe memory impairment), emotional changes (e.g., depression, apathy and anxiety), sleep perturbations (e.g., insomnia/hypersomnia), autonomic dysfunction (e.g., bladder disturbances, orthostatic hypotension, sweating), sensory symptoms (e.g., pain, visual and olfactory deficits) and gastrointestinal symptoms (e.g., constipation, nausea).

Parkinson's disease current treatment of choice is replacement of dopamine with its precursor Levodopa (L-Dopa), which unfortunately loses its effectiveness and can cause dyskinesia following prolonged usage. This fact motivates the search for new pharmacological strategies to better control the symptoms and/or progression of the disease.

The inverse relationship between smoking and PD has been confirmed by a number of epidemiological studies. Moreover, numerous preclinical studies indicate neuroprotective effects of nicotine. Thus, nicotine may offer a novel intervention in PD. Although use of nicotine patch has been suggested in some neurodegenerative disorders, including PD, the investigators believe that the key for success with nicotinic intervention, particularly in PD, relies on mode of nicotine administration. In our opinion, an optimal nicotinic therapy in PD would consist of pulsatile nicotine delivery (e.g. via nasal spray) similar to pulsatile nicotine obtained via smoking. Pulsatile stimulation of the central nicotinic receptors (achievable via nasal spray) would affect the dynamic of the nicotinic receptors much more desirably than continuous nicotine administration via patch, which can result in continuous nicotinic receptor desensitization. The investigators also believe that nicotine delivered via nasal spray, in addition to its potential usefulness for improving motor dysfunctions, may also be helpful in non-motor symptoms (e.g. cognitive decline and depression) that are commonly associated with neurological disorders such as PD.

Thus, this pilot clinical trial seeks to evaluate the efficacy of treatment during one month with nicotine nasal spray (Nicotrol NS®) in motor and non-motor aspects of PD.

Hypothesis: Scores of the Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) for motor and non-motor symptomatology will decrease after 1 month of treatment with nicotine nasal spray (Nicotrol) in patients with PD (stages 2-3 of Hoehn & Yahr).

Research question: Can controlled doses of nicotine administered via nasal spray decrease the severity of PD (stages 2-3 of Hoehn & Yahr) using MDS-UPDRS scores?

ELIGIBILITY:
Inclusion criteria:

* Subjects over 60 years of age with a clinical diagnosis of Parkinson's disease
* Stages of the disease 2-3 of Hoehn and Yahr
* Not exposed to tobacco during any stage of their life
* No history of lung diseases
* No laboratory abnormalities
* No history of adverse reactions to nicotine
* Able to use nicotine nasal spray
* Residents of Mexico City able to attend for evaluations
* Under current treatment with levodopa at a stable dose
* Not currently receiving a monoamine oxidase inhibitor treatment

Exclusion Criteria

* Unable to complete follow-up protocol
* Drug adverse reaction
* Death

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
Change from in motor dysfunction as assessed by MDS-UPDRS (Movement Disorder Society Unified Parkinson Disease subscale 3, range 0 best -56 worse ). | 1 month
  Change from baseline in motor dysfunction as assessed by MDS-UPDRS (Movement Disorder Society Unified Parkinson Disease subscale 3, range 0 best -56 worse ).

CONTACTS AND LOCATIONS:
Overall Officials: Mayela Rodríguez Violante, MSc., Principal Investigator — El Instituto Nacional de Neurologia Manuel Velasco Suarez
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía MVS, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Quik M. Smoking, nicotine and Parkinson's disease. Trends Neurosci. 2004 Sep;27(9):561-8. doi: 10.1016/j.tins.2004.06.008. PMID 15331239
- [Result] Tizabi Y, Getachew B. Nicotinic Receptor Intervention in Parkinson's Disease: Future Directions. Clin Pharmacol Transl Med. 2017;1(1):14-19. Epub 2017 Mar 6. PMID 29863173
- [Result] Tizabi Y, Getachew B, Rezvani AH, Hauser SR, Overstreet DH. Antidepressant-like effects of nicotine and reduced nicotinic receptor binding in the Fawn-Hooded rat, an animal model of co-morbid depression and alcoholism. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Apr 30;33(3):398-402. doi: 10.1016/j.pnpbp.2008.09.010. Epub 2008 Sep 19. PMID 18835320
- [Result] Villafane G, Cesaro P, Rialland A, Baloul S, Azimi S, Bourdet C, Le Houezec J, Macquin-Mavier I, Maison P. Chronic high dose transdermal nicotine in Parkinson's disease: an open trial. Eur J Neurol. 2007 Dec;14(12):1313-6. doi: 10.1111/j.1468-1331.2007.01949.x. Epub 2007 Oct 17. PMID 17941858
- [Result] Villafane G, Thiriez C, Audureau E, Straczek C, Kerschen P, Cormier-Dequaire F, Van Der Gucht A, Gurruchaga JM, Quere-Carne M, Evangelista E, Paul M, Defer G, Damier P, Remy P, Itti E, Fenelon G. High-dose transdermal nicotine in Parkinson's disease patients: a randomized, open-label, blinded-endpoint evaluation phase 2 study. Eur J Neurol. 2018 Jan;25(1):120-127. doi: 10.1111/ene.13474. Epub 2017 Oct 23. PMID 28960663